CLINICAL TRIAL: NCT01027676
Title: Phase I/II Study of Vorinostat and Gefitinib in Relapsed/ or Refractory Patients With Advanced Non-small Cell Carcinoma (NSCLC)
Brief Title: Study of Vorinostat and Gefitinib in Relapsed/ or Refractory Patients With Advanced Non-small Cell Carcinoma (NSCLC)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Ji-youn Han, Head, Center for Lung Cancer, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-09-433
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: Gefitinib; Vorinostat
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- study arm (Experimental): single arm Gefitinib plus vorinostat
  Interventions: Drug: Study treatment

INTERVENTIONS:
Drug: Study treatment — Gefitinib 250mg/QD plus vorinostat D1~7 & D15-21 / QD q 4weeks

SUMMARY:
Gefitinib is an orally active epidermal growth factor receptor-tyrosine kinase inhibitor (EGFR-TKI) and produces 8-20% of response rates in patients with advanced non-small cell lung cancer (NSCLC). Vorinostat (suberoylanilide hydroxamic acid [SAHA]) is a small-molecule inhibitor of histone deacetylase (HDAC) and induces cell differentiation, cell cycle arrest, and apoptosis in several tumor cells. There is a strong synergistic antiproliferative effect of vorinostat in combination with gefitinib in NSCLC cells. Vorinostat increases expression of E-cadherin and ErbB-3, which results in increased sensitivity to gefitinib. Moreover, In-vitro studies have shown that vorinostat leads to acetylation and disruption of Hsp90, which may lead to decreases in activity of pro-growth and prosurvival client proteins (J Bio Chem 2005;280:26729, Br J Cancer 2006;95:S2). These findings suggest that combination of vorinostat with gefitinib may improve the efficacy of gefitinib in NSCLC.

DETAILED DESCRIPTION:
Phase I design

* Three patients will be treated per cohort for one cycle (28 days per cycle).
* If no DLTs are recorded, treatment will continue and three patients will be treated in the subsequent cohort.
* However, if a patient develops a DLT, another three patients will be treated in this cohort for one cycle.
* If there are no more DLTs, dose escalation continues.
* If more than one of three patients develop a DLT in any cohort, another three patients will be treated in the next lower dosage cohort.
* If no DLTs are recorded in any of the cohorts, cohort 3 will be expanded to six patients.
* Up to 12 patients will be enrolled at the MTD.
* The phase II dose for this combined treatment will be therefore defined as the highest dosage cohort in which six patients had been treated and there are less than three DLTs.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of NSCLC, Stage IV or selected stage IIIB (with positive pleural effusion or multiple ipsilateral lung nodules) according to the American Joint Committee on Cancer (AJCC).
* Previously treated with at least one platinum-based chemotherapy.
* Before study entry, a minimum of 28 days must have elapsed since any prior chemotherapy.
* Prior radiation therapy is allowed as long as the irradiated area is not the only source of measurable disease.
* No other forms of cancer therapy, such as radiation, immunotherapy for at least 2 weeks before the enrollment in study.
* Performance status of 0-2 on the ECOG criteria.
* At least one unidimensionally measurable lesion meeting Response Evaluation Criteria in Solid Tumors (Revised RECIST guideline version 1.1)
* Estimated life expectancy of at least 8 weeks.
* Patient compliance that allow adequate follow-up.
* Adequate hematologic (WBC count 4,000/mm3, platelet count 150,000/mm3), hepatic (bilirubin level 1.5 mg/dL, AST/ALT 80 IU/L), and renal (creatinine concentration 1.5 mg/dL) function.
* Informed consent from patient or patient's relative.
* Males or females at least 18 years of age.
* If female: childbearing potential either terminated by surgery, radiation, or menopause, or attenuated by use of an approved contraceptive method (intrauterine device [IUD], birth control pills, or barrier device) during and for 3 months after trial. If male, use of an approved contraceptive method during the study and 3 months afterwards. Females with childbearing potential must have a urine negative hCG test within 7 days prior to the study enrollment.
* Patients with brain metastasis are allowed unless there were clinically significant neurological symptoms or signs

Exclusion Criteria:

* Presence of small-cell lung cancer alone or with NSCLC
* Unresolved chronic toxic effects from previous anticancer therapy: but patient could be enrolled, if they have recovered from any treatment-related toxicities NCI CTCAE grade ≤2
* Inability to swallow tablets
* Second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin or prior malignancy treated more than 5 years ago without recurrence).
* More than three previous chemotherapy regimens for NSCLC
* Previous treatment with any EGFR-TKI
* Patients who have been exposed to any prior HDAC inhibitor, with the exception of exception of valpronic acid used for treating seizures, provided there is a 30-day washout period
* Patients with active HIV or hepatitis B or C infection
* Concomitant use of phenytoin, carbamazepine, rifampicin, barbiturates, cyclosporine A, valpronic acid, Phenobarbital, ketoconazole, coumarin-derivative anticoagulants or St John's wort; severe or uncontrolled systemic disease; clinically active interstitial lung disease (except uncomplicated lymphangitic carcinomatosis) pregnancy; and breastfeeding.
* MI within preceding 6 months or symptomatic heart disease, including unstable angina, congestive heart failure or uncontrolled arrhythmia
* Serious concomitant infection including postobstructive pneumonia
* Major surgery other than biopsy within the past two weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-06; Primary Completion 2013-12 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | every 8 weeks
  The first day of treatment to the date that disease progression is reported or death date

SECONDARY OUTCOMES:
Overall Survival | every 8 weeks
  The first day of treatment to the date that death is reported or last survival status reported or
Objective Response rate | every 8 weeks
  The date of first evaluation to the date of disease progression

CONTACTS AND LOCATIONS:
Overall Officials: JI-YOUN HAN, M.D., Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Han JY, Lee SH, Lee GK, Yun T, Lee YJ, Hwang KH, Kim JY, Kim HT. Phase I/II study of gefitinib (Iressa((R))) and vorinostat (IVORI) in previously treated patients with advanced non-small cell lung cancer. Cancer Chemother Pharmacol. 2015 Mar;75(3):475-83. doi: 10.1007/s00280-014-2664-9. Epub 2015 Jan 1. PMID 25552401